CLINICAL TRIAL: NCT06491979
Title: Interventional Study on the Treatment of Uveitis With Vitamin and Unsaturated Fatty Acid Combination Dietary Supplements Through Modulating T Cell Function
Brief Title: Vitamin and Unsaturated Fatty Acid Supplements in Healthy and Uveitis Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Xiaomin Zhang, Principal Investigator, MD, PhD, Tianjin Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023KY-54
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Uveitis; Autoimmune Diseases
MeSH Terms: conditions — Uveitis; Autoimmune Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin A treatment (Experimental)
  Interventions: Dietary Supplement: Vitamin A treatment
- Monounsaturated fatty acid mixture (Experimental)
  Interventions: Dietary Supplement: Monounsaturated fatty acid mixture
- Polyunsaturated fatty acid mixture (Experimental)
  Interventions: Dietary Supplement: Polyunsaturated fatty acid mixture
- Fatty acid mixture (Experimental)
  Interventions: Dietary Supplement: Fatty acid mixture

INTERVENTIONS:
Dietary Supplement: Vitamin A treatment — Vitamin A, 32 microgram per kilograms (of body weight) per day, for three weeks
  Arms: Vitamin A treatment
Dietary Supplement: Monounsaturated fatty acid mixture — Monounsaturated fatty acid mixture (mainly Omega-7, Omega-9), 47 milligrams per kilogram (of body weight) per day, for three weeks
  Arms: Monounsaturated fatty acid mixture
Dietary Supplement: Polyunsaturated fatty acid mixture — Polyunsaturated fatty acid mixture (mainly Omega-3, Omega-6), 6 milligrams per kilogram (of body weight) per day, for three weeks
  Arms: Polyunsaturated fatty acid mixture
Dietary Supplement: Fatty acid mixture — Fatty acid mixture (mainly saturated fatty acid, Omega-6, Omega-7, Omega-9), 83 milligrams per kilogram (of body weight) per day, for three weeks
  Arms: Fatty acid mixture

SUMMARY:
The goal of this clinical trial is to learn if dietary supplements containing vitamin and unsaturated fatty acid works to intervene T cell inflammatory factor expression in patients with uveitis and healthy subjects in adults.

ELIGIBILITY:
Inclusion Criteria:

* healthy or with uveitis volunteers age 19-65 years.

Exclusion Criteria:

* abnormal blood glucose, blood pressure, blood lipids, or other systemic diseases should not participate in the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory factors-Interleukin-17A (IL-17A) | 3 weeks
  Flow cytometry analysis of peripheral blood mononuclear cells (PBMCs) to detect the ratio of Interleukin-17A (IL-17A) -producing cells in CD4+ T cells and CD8+ T cells
Inflammatory factors-Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) | 3 weeks
  Flow cytometry analysis of peripheral blood mononuclear cells (PBMCs) to detect the ratio of Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) -producing cells in CD4+ T cells and CD8+ T cells
Inflammatory factors-Interferon gamma (IFN-γ) | 3 weeks
  Flow cytometry analysis of peripheral blood mononuclear cells (PBMCs) to detect the ratio of Interferon gamma (IFN-γ) -producing cells in CD4+ T cells and CD8+ T cells

SECONDARY OUTCOMES:
Cytokine levels-Interleukin-17A (IL-17A) | 3 weeks
  Analysis of cytokine levels in blood. Detect the concention of Interleukin-17A (IL-17A) in plasma
Cytokine levels-Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) | 3 weeks
  Analysis of cytokine levels in blood. Detect the concention of Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) in plasma
Cytokine levels-Interferon gamma (IFN-γ) | 3 weeks
  Analysis of cytokine levels in blood. Detect the concention of Interferon gamma (IFN-γ) in plasma
Cytokine levels-Interleukin-2 (IL-2) | 3 weeks
  Analysis of cytokine levels in blood. Detect the concention of Interleukin-2 (IL-2) in plasma
Cytokine levels-Interleukin-10 (IL-10) | 3 weeks
  Analysis of cytokine levels in blood. Detect the concention of Interleukin-10 (IL-10) in plasma
Cytokine levels-Interleukin-9 (IL-9) | 3 weeks
  Analysis of cytokine levels in blood. Detect the concention of Interleukin-9 (IL-9) in plasma
Cytokine levels-Interleukin-4 (IL-4) | 3 weeks
  Analysis of cytokine levels in blood. Detect the concention of Interleukin-4 (IL-4) in plasma
Cytokine levels-Tumor Necrosis Factor alpha (TNF-α) | 3 weeks
  Analysis of cytokine levels in blood. Detect the concention of Tumor Necrosis Factor alpha (TNF-α) in plasma

OTHER OUTCOMES:
Transcriptomics analysis | 3 weeks
  Analyze the changes in peripheral blood mononuclear cells using transcriptomics. Detect the cell populations , genes number and expression.
Proteomics analysis | 3 weeks
  Analyze the changes in peripheral blood mononuclear cells using proteomics. Detect the proteins expression.
post-translational modification proteomics analysis | 3 weeks
  Analyze the changes in peripheral blood mononuclear cells using post-translational modification proteomics. Detect the protein various modification, such as lactylation, crotonylation, palmitoylation and methylation.
metabolomics analysis | 3 weeks
  Analyze the changes in peripheral blood mononuclear cells using metabolomics. Detect the metabolites numbers, localization and level.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China